CLINICAL TRIAL: NCT04557514
Title: Comparative Study Between Fat Injection And Platelet Rich Plasma IN Post Burn Facial Scar Clinical And Histopathological Assessment
Brief Title: Comparative Study Between Fat Injection And Platelet Rich Plasma In Post Burn Facial Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mostafa Shehata Mohammed, official investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: facial burn scar
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Burn Scar
MeSH Terms: interventions — CD36 Antigens

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich plasma injection in post burn facial scar (Active Comparator): prp in subgroup allocation 1:1 Obtain WB by venipuncture in acid citrate dextrose (ACD) tubes
  Do not chill the blood at any time before or during platelet separation.
  Centrifuge the blood using a 'soft' spin.
  Transfer the supernatant plasma containing platelets into another sterile tube (without anticoagulant).
  Centrifuge tube at a higher speed (a hard spin) to obtain a platelet concentrate.
  The lower 1/3rd is PRP and upper 2/3rd is platelet-poor plasma (PPP). At the bottom of the tube, platelet pellets are formed.
  Remove PPP and suspend the platelet pellets in a minimum quantity of plasma (2-4 mL) by gently shaking the tube.
  Interventions: Procedure: platelet rich plasma injection in post burn facial scar; Procedure: fat injection in post burn facial scar
- fat injection in post burn facial scar (Active Comparator): After aspiration of the fatty tissue, it is important that nonviable components of the aspirate, such as oil, blood, and local anesthetics are removed and, at the same time, the quality, integrity, and viability of the adipocytes and the inherent mesenchymal stem cells in the aspirate be maintained. Processing techniques are sedimentation , filtering and washing There is no consensus as to the optimal method of fat graft preparation.
  Interventions: Procedure: platelet rich plasma injection in post burn facial scar; Procedure: fat injection in post burn facial scar

INTERVENTIONS:
Procedure: platelet rich plasma injection in post burn facial scar — 2 spins>>>
  1. st spin (separate plasma from blood) 2500 for 10 minutes
  2. nd spin (separate platelet rich part of plasma) 1500 for 10 minutes Taking lower part (platelet rich plasma ) Injection under scar after rigotomy
Procedure: fat injection in post burn facial scar — Anesthesia : general or local Lipoaspirate from abdomen or thigh using adrenaline(1\1000000) + ringer lactate + zylocaine Liposuction by canula no4 Sediment 3 layers : taking mid layer of fat and omit uppermost and lowermost layers Lipoinjection in fan shaped manner 10-20 cc according to site affected by canula no 1 .

SUMMARY:
Best method in management of facial burn scar

DETAILED DESCRIPTION:
The stages of wound healing:proceed in an organized way and follow four processes: hemostasis, inflammation, proliferation and maturation. Although the stages of wound healing are linear, wounds can progress backward or forward depending on internal and external patient conditions. The four stages of wound healing are:Hemostasis Phase Hemostasis is the process of the wound being closed by clotting. Hemostasis starts when blood leaks out of the body. Inflammatory Phase Inflammation is the second stage of wound healing and begins right after the injury when the injured blood vessels leak transudate (made of water, salt, and protein) causing localized swelling. Proliferative Phase The proliferative phase of wound healing is when the wound is rebuilt with new tissue made up of collagen and extracellular matrix. Maturation Phase Also called the remodeling stage of wound healing, the maturation phase is when collagen is remodeled from type III to type I and the wound fully closes.

Fat Injection In Facial burn scar:The effects of the lipofilling can be seen starting from 3 weeks after the procedure, in terms of better scar color, pliability, thickness, relief, itching, pain, scar vascularization and pigmentation. Indeed, autologous fat grafting makes the skin softer, more flexible and extensible; besides, the color seems similar to the surrounding unharmed skin.

Platelet Rich Plasma In Facial burn scar: Impaired wound-healing and a long treatment course in severe burns as well as secondary complications originating from uncovered wounds motivate research to accelerate the wound-healing process and speed up re-epithelialization in burn patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients With Post Burn Facial Scar
2. Age: 15 _60 Yrs Old
3. Mature Burn Scar (After 3 Months)

Exclusion Criteria:

1. Patients Less Than 15 Yrs Old
2. Patients More Than 60 Yrs Old
3. Patients With Comorbidies (Hypertension-Diabetes-Thromboembolic Diseases-Immunocomprimized Patients)
4. Patients With Burn Scar In Any Site Of Body Other Than Face

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
vancouver scale | 3 months
  Pigmentation (0-2) Normal 0 Hypopigmentation 1 Hyperpigmentation 2 Vascularity (0-3) Normal 0 Pink 1 Red 2 Purple 3 Pliability (0-5) Normal 0 Supple 1 Yielding 2 Firm 3 Banding 4 Contracture 5 Height (0-3) Normal (flat) 0 0-2 mm 1 2-5 mm 2 >5 mm 3

CONTACTS AND LOCATIONS:
Overall Officials: wagdi mohamed, lecturer, Study Director — lecturer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhooshan LS, Devi MG, Aniraj R, Binod P, Lekshmi M. Autologous emulsified fat injection for rejuvenation of scars: A prospective observational study. Indian J Plast Surg. 2018 Jan-Apr;51(1):77-83. doi: 10.4103/ijps.IJPS_86_17. PMID 29928084
- [Background] Ozcelik U, Ekici Y, Bircan HY, Aydogan C, Turkoglu S, Ozen O, Moray G, Haberal M. Effect of Topical Platelet-Rich Plasma on Burn Healing After Partial-Thickness Burn Injury. Med Sci Monit. 2016 Jun 5;22:1903-9. doi: 10.12659/msm.895395. PMID 27262706